CLINICAL TRIAL: NCT06786234
Title: An Open-Label, Phase 1b Study to Evaluate Safety, Tolerability & Preliminary Activity of the CTPS1 Inhibitor STP938 in Adult Subjects With High Risk Essential Thrombocythaemia Who Are Resistant to or Intolerant of Hydroxycarbamide Therapy
Brief Title: A Phase 1 Study to Assess STP938 as a Monotherapy in Adults With High Risk Essential Thrombocythaemia
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Step Pharma, SAS (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STP938-301
Record Dates: First submitted 2025-01-08; First posted 2025-01-22 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Essential Thrombocythaemia
Keywords: Essential Thrombocythemia; High risk; Resistant to or Intolerant of Hydroxycarbamide Therapy; Resistant to or Intolerant of Hydroxyurea Therapy; Oral therapy
MeSH Terms: conditions — Thrombocythemia, Essential

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Phase 1b (Experimental): Up to 5 dose levels with STP938 administered as oral therapy
  Interventions: Drug: STP938

INTERVENTIONS:
Drug: STP938 — At enrolment all patients will be assigned to a single dose level of STP938 for 4 weeks. After 4 weeks the dose level may be adjusted as needed by the Investigator.

SUMMARY:
The goal of this clinical trial is to learn if the drug STP938 works to treat adults with high risk essential thrombocythaemia (ET) who are resistant to, or intolerant of, hydroxycarbamide (also known as hydroxyurea) therapy. The trial will also learn about the safety of STP938. The main questions the trial aims to answer are:

* Does STP938 control platelet counts
* Does STP938 control platelet counts without inducing unwanted side effects

Participants will:

* Take STP938 every day for up to 12 months.
* Visit the clinic once every week for the first month, then every 2 weeks for checkups and tests.
* Complete a questionnaire about symptoms once a month.

DETAILED DESCRIPTION:
The aim of the study is to assess a new drug called STP938 for the treatment of essential thrombocythaemia (ET). The study with assess how effective STP938 in treating ET, and also assess any side effects of taking the drug. The study will enrol individuals with high risk ET who require treatment to lower their platelet count. Individuals enrolling on the study will have already tried treatment with hydroxycarbamide (also known as hydroxyurea) but are in need of a different treatment as hydroxycarbamide either did not control the platelet count or produced unwanted side effects.

STP938 is a new class of drug that inhibits the enzyme cytidine triphosphate synthase 1 (CTPS1). Inhibition of CTPS1 is a novel way of lowering the platelet count. This study is a phase 1b, open-label, multicentre trial. Participants will receive STP938 capsules every day, in cycles of 28 days, for approximately 12 months. Participants may continue to receive study drug for a longer period, so long as it is controlling the platelet count and not causing side effects. During the study, participants will visit the study site about 26 times (2 times per cycle) over an estimated 12 months. Once the treatment is complete, safety follow-up visit(s) will occur to make sure the participant is not experiencing any adverse effects. The following study procedures will be performed: (a) physical examinations (b) ECGs (c) blood tests, (d) urine tests (e) CT/MRI scans (f) bone marrow biopsies (g) drug administration (h) study drug blood level tests and (i) gene testing.

ELIGIBILITY:
Key Inclusion Criteria:

* Adults aged 18 years or older
* A confirmed diagnosis of ET according to World Health Organisation (WHO) or British Society for Haematology (BSH) criteria.
* Meeting criteria for high risk ET.
* Raised platelet count (>600 x109/L) requiring cytoreductive therapy.
* Neutrophil count >1.0 x109/L.
* Either intolerant of or resistant to hydroxycarbamide having met any one of the criteria at any point in their disease whilst receiving hydroxycarbamide.
* Adequate hepatic function.
* Adequate blood coagulation parameters.
* Eastern Cooperative Oncology Group (ECOG) status of 0-2.

Key Exclusion Criteria:

* Subjects currently or recently receiving cytoreductive therapy for the treatment of essential thrombocythaemia (wash out periods apply).
* Subjects who have received any investigational agents for the treatment of essential thrombocythaemia within 4 weeks before enrolment or less than 5 half-lives since completion of prior therapy, whichever is shorter.
* Proven or suspected transformation to polycythaemia vera, myelofibrosis, myelodysplasia, acute myeloid leukaemia or another myeloid neoplasm.
* Known malabsorption syndrome or other condition that may impair absorption of study medication (e.g. gastrectomy).
* Previous splenectomy.
* Any uncontrolled intercurrent illness.
* Immunocompromised subjects with increased risk of opportunistic infections.
* Known active or chronic hepatitis B or active hepatitis C virus (HCV) infection.
* Pregnant females, breastfeeding females, and women of child bearing age or males not willing to comply with contraceptive requirements.
* Known hypersensitivity to any of the excipients used in the formulation of the study drug.
* Corrected QT interval >470 msec based on averaged triplicate electrocardiogram (ECG) readings at the Screening Visit using the QT interval corrected for heart rate using Fridericia's method (QTcF).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-06-18 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Clinical Efficacy | Through study completion, an average of 12 months
  Complete and partial response rates per European LeukemiaNet criteria
Safety and Tolerability | Through study completion, an average of 12 months
  Toxicity profile based on National Cancer Institute Common Terminology Criteria for Adverse Events

SECONDARY OUTCOMES:
Durability of Response to STP938 | Through study completion, an average of 12 months
  Time from achieving response to loss of response
Impact of STP938 on Disease-Related Complications | Through study completion, an average of 12 months
  Prevalence of haemorrhagic complications, thromboembolic events and disease transformation.

OTHER OUTCOMES:
Patient Reported Outcomes and Symptom Burden | Through study completion, an average of 12 months
  Myeloproliferative Neoplasm Symptom Assessment Form (18 item). Minimum value is zero (0); the maximum value is 180. A score of zero equates to absence of symptoms, higher scores equate to worse outcome.
Molecular Response | Through study completion, an average of 12 months
  Change in Variant Allele Fraction: For known ET-associated mutations.
Bone Marrow Histology | Screening and Cycle 12 (each cycle is 28 days)
  Changes in Histological Appearances
Spleen Volume | Through study completion, an average of 12 months
  Change in Spleen Volume: Measured by MRI or CT scan.

CONTACTS AND LOCATIONS:
Overall Officials: Maureen Higgins, Study Director — Step Pharma
Locations (13):
- France (7):
  - CHU Brest, Brest
  - Institut Paoli-Calmettes, Marseille
  - CHU Nantes, Nantes
  - CHU Nice, Nice
  - CHU Nîmes, Nîmes
  - Hôpital Saint-Louis, Paris
  - Gustave Roussy, Villejuif
- United Kingdom (6):
  - Royal Hallamshire Hospital, Sheffield, South Yorkshire
  - University Hospital of Wales, Cardiff
  - Imperial College London / Hammersmith Hospital, London
  - Sarah Cannon Research Institute, London
  - Cancer and Haematology Centre, Churchill Hospital, Oxford
  - University of Southampton Hospital, Southampton

IPD SHARING:
Plan to Share IPD: No